CLINICAL TRIAL: NCT03403530
Title: A Prospective Study to Analyze the Efficacy of IgM Rich Immunoglobulin as an Adjunct to Antibiotics in the Treatment of Bacterial Sepsis in Very Low Birth Weight Preterm Neonates
Brief Title: Efficacy of IgM Rich Immunoglobulin With Antibiotics for Bacterial Sepsis in Very Low Birth Weight Preterm Neonates
Acronym: IgMNS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Takhtasinhji General Hospital (Other Government)
Responsible Party: Principal Investigator, Sonal V Jindal, Principal Investigator, Resident, Sir Takhtasinhji General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: svjindal
Record Dates: First submitted 2018-01-01; First posted 2018-01-18 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Neonatal SEPSIS; Very Low Birth Weight Baby
Keywords: IgM; Immunoglobulin; Neonatal sepsis; very low birth weight preterm
MeSH Terms: conditions — Neonatal Sepsis | interventions — pentaglobulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- case group (Active Comparator): 'IgM rich immunoglobulin' intravenous infusion in the dose of 5 ml/ kg/ dose over 3 hours once a day for 3 days.
  Interventions: Drug: IgM rich Immunoglobin
- control group (Placebo Comparator): antibiotics only
  Interventions: Drug: IgM rich Immunoglobin

INTERVENTIONS:
Drug: IgM rich Immunoglobin — the 'IgM rich immunoglobn' is the normal human immunoglobin containing Human plasma protein 50mg/ml of which immunoglobin is atleast 95% Immunoglobin M (IgM) 6mg Immunoglobin A (IgA) 6mg Immunoglobin G (IgG) 38mg
  Other Names: Pentaglobin®

SUMMARY:
Study comprises of giving IVIG to half of the septic VLBW preterm neonates along with ongoing antibiotics and placebo to the other half. The immunoglobulin will be given for 3 days and neonates will be monitored for the results. The data will be analysed on the basis of blood culture results and outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Preterm
* Very low birth weight baby: birth weight 1-1.5 kg
* Both inside and outside delivered babies
* Gender: males and females
* Probable severe sepsis (septic score)

Exclusion Criteria:

* Extremely low birth weight babies: < 1 kg
* Babies >1.5 kg birth weight
* Babies born with congenital malformations
* Full term babies
* IUGR babies
* Child with no signs of sepsis
* HBsAg Positive
* HIV Positive

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Discharge rates | 6 months
  patients who received IgM rich Immunoglobin along with antibiotics have better outcome as compared to the patients who receive only antibiotics.

SECONDARY OUTCOMES:
Duration of hospital stay | 6 months
  patients who received IgM rich Immunoglobin along with antibiotics have better outcome as compared to the patients who receive only antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Jayendra R Gohil, MD, Principal Investigator — SirTakhtasinhjiGH, Prof Pediatrics, Govt MC, Bhavnagar
Locations (1):
- NICU, Sir T Hospital, Bhavnagar, Bhavnagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Capasso L, Borrelli A, Cerullo J, Pisanti R, Figliuolo C, Izzo F, Paccone M, Ferrara T, Lama S, Raimondi F. Role of immunoglobulins in neonatal sepsis. Transl Med UniSa. 2014 Dec 19;11:28-33. eCollection 2015 Jan-Apr. PMID 25674546
- [Result] Haque KN, Zaidi MH, Bahakim H. IgM-enriched intravenous immunoglobulin therapy in neonatal sepsis. Am J Dis Child. 1988 Dec;142(12):1293-6. doi: 10.1001/archpedi.1988.02150120047038. PMID 3195529